CLINICAL TRIAL: NCT00819299
Title: A Prospective, Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the AcuFocus Corneal Inlay (ACI)™ ACI 7000PDT in Presbyopic Subjects
Brief Title: Safety and Effectiveness Study of the AcuFocus Corneal Inlay ACI 7000PDT in Presbyopes
Acronym: ACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACU-P08-020
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Presbyopia
Keywords: Presbyopia; accommodation; near visual acuity; LASIK
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AcuFocus Corneal Inlay (Experimental): Implantation of the AcuFocus Corneal Inlay ACI 7000PDT in emmetropic presbyopic patients.
  Interventions: Device: AcuFocus Corneal Inlay ACI 7000PDT

INTERVENTIONS:
Device: AcuFocus Corneal Inlay ACI 7000PDT — corneal inlay
  Other Names: AcuFocus KAMRA inlay

SUMMARY:
The purpose of this study is to determine if the AcuFocus Corneal Inlay ACI 7000PDT will provide an effective method for the correction of presbyopia in patients who have normal distance vision but need a correction such as glasses or contact lenses to see clearly at near.

DETAILED DESCRIPTION:
The loss of near vision and the ability to perform tasks that require near vision is part of the normal aging process. This natural transformation in the eye occurs as a result of the loss of accommodation of the crystalline lens, a condition known as presbyopia. The crystalline lens is responsible for the accommodative properties of the human eye, as established by Young in 1801, over 200 years ago.1 During accommodation, the ciliary muscle contracts, decreasing tension on the zonules, and allowing the crystalline lens to thicken, increasing its refractive power. This mechanism of accommodation and thickening of the lens provides the eye with adequate refractive power for near vision. The loss of accommodation with aging is the result of changes in the crystalline lens composition that prevent the natural accommodative process from occurring. This is associated with the gradual loss of near vision without external correction, generally in the form of spectacles.

The AcuFocus™ ACI 7000PDT represents new technology based on the well-established concept of small-aperture optics. In early cameras, depth of focus was controlled by reducing the aperture through which light enters. The smaller the aperture, the greater the depth of focus will be. This concept also applies to the human eye. In the eye of a presbyopic emmetrope, the lens cannot accommodate sufficiently to focus the light rays from a near object onto a single point on the retina. Thus, a point object is imaged as a blur circle on the retina, and images of extended objects are degraded as well. If an opaque disc with a small aperture in the center is placed in front of the eye, the peripheral rays will be obscured while the central rays pass unaffected. Since peripheral rays enter the eye at a larger angle, they create a larger blur circle at the retinal image plane. Eliminating these peripheral rays reduces the size of the blur circle, improving image resolution.

In presbyopic subjects, objects closer than arm's length are focused behind the retina, thus creating blurred retinal images (which are composed of blur circles). A small aperture inlay placed in front of the eye of these subjects allows them to see at near by reducing the size of the blur circle.

AcuFocus, Inc. has developed a stationary intracorneal inlay designed to create a small aperture effect. The implant is intended to be placed intra-stromally; the corneal flap will be newly created and fully lifted for presbyopic emmetropes. Placement of the ACI on the stromal bed centered over the pupil in the non-dominant eye is expected to increase the depth of focus of the eye by reducing the circle of blur. Based on theoretical calculations of small aperture optics, the ACI is expected to provide presbyopic subjects with improvement of near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be natural emmetropes needing a minimum magnitude of +1.00D to +2.50D of reading add.
2. Subjects must have uncorrected near visual acuity worse than 20/40 and better than 20/100 in the eye to be implanted.
3. Subject must have distance visual acuity correctable to at least 20/20 in both eyes.
4. Subjects must have a preoperative spherical equivalent of plano defined as +0.50D to -0.75D with no more than 0.75D of refractive cylinder as determined by cycloplegic refraction in the eye to be implanted.

Exclusion Criteria:

1. Subjects with a difference of > 1.00D between the spherical equivalent manifest refraction and the spherical equivalent cycloplegic refraction.
2. Subjects with anterior segment pathology, including cataracts, in the eye to be implanted.
3. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormalities (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in the eye to be implanted.
4. Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in the eye to be implanted.
5. Subjects with a history of chronic dry eye not responding to therapy.
6. Subjects with distorted or unclear corneal mires on topography maps of the eye to be implanted.
7. Subjects who require canthotomy to generate a corneal flap in the eye to be implanted.
8. Subjects with macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in the eye to be implanted.
9. Subjects who have undergone previous intraocular or corneal surgery including cataract and LASIK surgery.
10. Subjects with a history of herpes zoster or herpes simplex keratitis.
11. Subjects who have a history of steroid-responsive rise in intraocular pressure, preoperative IOP > 21 mmHg, glaucoma, or is a glaucoma suspect.
12. Subjects with a history of diagnosed diabetes, autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
13. Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immunocompromised subjects.
14. Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of any ocular pathology including ocular allergy.
15. Subjects using systemic medications with significant ocular side effects.
16. Subjects who are pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
17. Subjects with known sensitivity to planned study concomitant medications.
18. Subjects who are participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 359 (Actual)
Dates: Start 2008-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improvement in uncorrected near visual acuity | 12 months
  Increased depth of focus created by the small aperture of the ACI to improve near visual acuity, while maintaining a range of focus over intermediate and distance.

SECONDARY OUTCOMES:
Subjective improvement in near visual acuity as measured by subjective questionnaire. | 12 months
  Questionnaire assessed 1) improvement in near vision 2) satisfaction with the outcome of procedure 3) near vision tasks for exploratory analysis 4) distance vision tasks for exploratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Perry Binder, MD, Study Director
Locations (15):
- United States (15):
  - McDonald Eye Associates, Fayetteville, Arkansas
  - Maloney Vision, Los Angeles, California
  - TLC Laser Eye Center, Newport Beach, California
  - Gordon Binder Weiss Vision Institute, San Diego, California
  - Eye Center NOCO, Fort Collins, Colorado
  - Kraff Eye Institute, Chicago, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Pepose Vision Institute, Chesterfield, Missouri
  - The Cornea & Laser Eye Institute, P.A, Teaneck, New Jersey
  - Coleman Vision, Albuquerque, New Mexico
  - University of Rochester Eye Institute - Strong Vision, Rochester, New York
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Hoopes Vision, Sandy City, Utah
  - Davis Duehr Dean, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website — http://www.acufocus.com